CLINICAL TRIAL: NCT05521269
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ANX1502 in Normal Healthy Volunteer
Brief Title: Dose Study of ANX1502 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Annexon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: ANX1502-NHV-01; 2022-000594-21 (EudraCT Number)
Record Dates: First submitted 2022-08-28; First posted 2022-08-30 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: healthy

STUDY DESIGN:
Intervention Model Description: This study consists of single-ascending dose (SAD), food effect, and multiple-ascending dose (MAD) parts.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANX1502 SAD (Experimental): Participants will be administrated a single oral dose of ANX1502 at various ascending dose levels or matching placebo.
  Interventions: Drug: ANX1502; Drug: Placebo
- ANX1502 MAD (Experimental): Participants will be administrated multiple oral doses of ANX1502 at various ascending dose levels or matching placebo for 14 days.
  Interventions: Drug: ANX1502; Drug: Placebo

INTERVENTIONS:
Drug: ANX1502 — ANX1502 is a prodrug of ANX1439.
Drug: Placebo — Placebo comparator.

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of ANX1502 (prodrug) and ANX1439 (active drug) in healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Must be healthy as determined by medical evaluation including medical history, physical examination, vital signs assessments (including supine blood pressure, supine pulse rate, respiration rate, and temporal body temperature), 12-lead electrocardiogram (ECG), and laboratory tests.
* MAD cohorts only: Documented history of vaccinations within 5 years of Screening or willing to undergo vaccinations prior to Screening against encapsulated bacterial pathogens.

Key Exclusion Criteria:

* History or presence of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, malabsorption syndrome, metabolism, or elimination of drugs; constituting a risk when taking the study drug; or interfering with the interpretation of data. Exceptions can be made for individuals with childhood or remote disorders that are no longer active.
* History of any autoimmune disease
* History of meningitis or septicemia
* Clinically significant infection within 30 days prior to study drug administration that required medical intervention
* Known genetic deficiencies of the complement cascade system or immunodeficiency.
* Clinically significant illness within 4 weeks of the start of dose administration as determined by the Investigator.
* Clinically significant multiple or severe drug allergies, or severe post-treatment hypersensitivity reactions .
* History of prior other malignancy that could affect compliance with the protocol or interpretation of results
* Has clinically significant laboratory abnormalities or abnormal ECG
* History of splenectomy.
* Antinuclear antibodies titer ≥1:160 at Screening.
* Has donated blood or plasma within 30 days prior to Screening or had a loss of whole blood of more than 500 milliliter (mL) within the 30 days prior to Screening, or receipt of a blood transfusion within one year prior to Screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) After A Single Dose and Multiple Doses of ANX1502 | Day 1 (after dosing) through Day 29

SECONDARY OUTCOMES:
Plasma ANX1502 and ANX1439 Concentrations After A Single Dose and Multiple Doses of ANX1502 | Predose up Day 29
Maximum Observed Plasma Concentration (Cmax) of ANX1502 and ANX1439 After A Single Dose and Multiple Doses of ANX1502 | Predose up Day 29
Observed Time to Cmax (Tmax) of ANX1502 and ANX1439 After A Single Dose and Multiple Doses of ANX1502 | Predose up to Day 29
Area Under the Concentration-time Curve (AUC) of ANX1502 and ANX1439 After A Single Dose and Multiple Doses of ANX1502 | Predose up Day 29
Terminal Half-life (t1/2) of ANX1502 and ANX1439 After A Single Dose and Multiple Doses of ANX1502 | Predose up to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Olga Bandman, Study Director — Annexon, Inc.
Locations (1):
- Annexon Investigational Site 01, Groningen, Netherlands